CLINICAL TRIAL: NCT05243849
Title: Characterization of Retinal Microvascular and FAZ Changes in Ischemic Stroke and Its Different Types
Status: Unknown | Type: Observational
Last Known Status: Recruiting
Sponsor: Peking University Third Hospital (Other)
Responsible Party: Sponsor
Other Study IDs: OCTA
Record Dates: First submitted 2021-12-29; First posted 2022-02-17 (Actual); Last update posted 2022-02-17 (Actual); Status verified 2021-12

CONDITIONS: Ischemic Stroke
Keywords: Ischemic Stroke; Optical Coherence Tomography Angiography; Retina
MeSH Terms: conditions — Ischemic Stroke

STUDY DESIGN:
Observational Model: Case-Control | Time Perspective: Cross-Sectional
Oversight: Data Monitoring Committee: Yes

GROUPS / COHORTS (2):
- Ischemic Stroke: The diagnosis of ischemic stroke was obtained from previous diagnostic reports or electronic medical records, according to the diagnostic criteria from the Trial of Org 10172 in Acute Stroke Treatment (TOAST).
  Interventions: Device: Optical Coherence Tomography Angiography
- Control: Inclusion criteria for healthy controls were no history of ischemic stroke or other neurological and ocular diseases.
  Interventions: Device: Optical Coherence Tomography Angiography

INTERVENTIONS:
Device: Optical Coherence Tomography Angiography — Optical coherence tomography angiography (OCTA) is a novel non-invasive, non-dye and high-resolution imaging technique, allowing real-time quantitative evaluation of retinal vasculature and the structure of foveal avascular zone (FAZ).

SUMMARY:
The study aimed to access the microvascular changes in the superficial capillary plexus (SCP) and deep capillary plexus (DCP) in patients with ischemic stroke and its different types using optical coherence tomography angiography.

DETAILED DESCRIPTION:
Investigators used OCTA to quantitatively access the retinal microvasculature of SCP and DCP, aiming to detect the geometry changes of retinal microvasculature and FAZ in ischemic stroke patients and its different types.

ELIGIBILITY:
Inclusion Criteria:

Patients who were diagnosed with ischemic stroke by MRI were scheduled for an OCTA examination. The diagnosis of ischemic stroke was obtained from previous diagnostic reports or electronic medical records, according to the diagnostic criteria from the Trial of Org 10172 in Acute Stroke Treatment (TOAST).

Exclusion Criteria:

1) Retinal diseases or diseases affecting vessel structure in fundus photography, including age-related maculopathy; diabetic retinopathy, central serous chorioretinopathy, retinal pigment epithelial detachment and glaucoma); poor cooperation in ophthalmic examinations; high refractive error (>+6.00 D or <-6.00 D Spherical Equivalent); low-quality OCTA images (signal strength index < 6/10). Inclusion criteria for healthy controls were no history of ischemic stroke or other neurological and ocular diseases.

Ages: 40 Years to 80 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Study Population: Patients who were diagnosed with ischemic stroke by MRI and healthy controls were scheduled for an OCTA examination.
Sampling Method: Non-Probability Sample
Enrollment: 100 (Estimated)
Dates: Start 2022-01-01 (Actual); Primary Completion 2022-06 (Estimated); Study Completion 2022-06 (Estimated)

PRIMARY OUTCOMES:
Vascular Area Density(VAD) | immediately after meeting the inclusion and exclusion criteria
  The total length in millimeters of perfused retinal microvasculature per unit area in square millimeters in the annular region of analyzed area
Vascular Fractal Dimension(VFD) | immediately after meeting the inclusion and exclusion criteria
  A well-known parameter which indicates the degree of geometric complexity of vasculature
Vascular Orientation Distribution(VOD) | immediately after meeting the inclusion and exclusion criteria
  The direction of each vascular pixel to indicate the trend of the blood flow
FAZ Area(FA) | immediately after meeting the inclusion and exclusion criteria
  The total numbers of pixels in the FAZ region
FAZ Axis Ratio(FAR) | immediately after meeting the inclusion and exclusion criteria
  The ratio between the major and minor axes of the fitted ellipse from the FAZ boundary. The axis ratio of a perfect circular FAZ is equal to 1
FAZ Circularity(FC) | After meeting the inclusion and exclusion criteria
  The ratio of the perimeter of the FAZ to the parameter of a circle with equal area, reflecting the degree of roundness of the FAZ
FAZ Roundness(FR) | immediately after meeting the inclusion and exclusion criteria
  Similar to FC, but is less sensitive to irregular borders along the parameter of FAZ

CONTACTS AND LOCATIONS:
Overall Officials: Hongyu Duan, MD, Study Director — Peking University Third Hospital
Locations (1):
- Peking University Third Hospital, Beijing, China

IPD SHARING:
Plan to Share IPD: No